CLINICAL TRIAL: NCT04901858
Title: Pilot Study Into the Structural Local Molecular Environment Following an ACL Injury
Brief Title: Knee Aspiration and High Definition MRI for ACL Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Responsible Party: Principal Investigator, Mr Stephen McDonnell, Principal Investigator, Cambridge University Hospitals NHS Foundation Trust
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: A095100
Record Dates: First submitted 2021-02-03; First posted 2021-05-26 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: ACL Injury
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Aspiration of haemarthrosis and high definition MRI — Aspiration of haemarthrosis and high definition MRI

SUMMARY:
The aim of this pilot study is to understand the biological changes that occur within the knee joint following injury to the anterior cruciate ligament (ACL). This will be achieved through aspiration and analysis of the haemarthrosis which fills the knee following injury. The study will look at inflammatory and healing responses using DNA, RNA and protein analysis.

This, combined with high resolution imaging of the knee and surrounding soft tissue structures, may enable a more patient specific approach to treatment of ACL injury.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of ACL injury confirmed by MRI
* All participants must have the capacity to provide informed consent to participate
* Participants must be able to comply with required study visit

Exclusion Criteria:

* Participants outside of the specified age range
* Participants who do not have the mental capacity to make informed decisions
* Participants who have meniscal pathology or other injuries requiring urgent surgery

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Estimated)
Dates: Start 2019-11-22 (Actual); Primary Completion 2024-11 (Estimated); Study Completion 2024-11 (Estimated)

PRIMARY OUTCOMES:
Pattern of injury on High Definition MRI measured by comparison with 3t MRI images | Last visit, usually 28 days
  Outcome will illustrate any additional benefit of high definition MRI

SECONDARY OUTCOMES:
Identification of acute inflammatory mediators measured by NanoString molecular analysis | Last visit, usually 28 days

CONTACTS AND LOCATIONS:
Locations (1):
- Cambridge University Hospitals NHS Foundation Trust, Cambridge, United Kingdom